CLINICAL TRIAL: NCT05884099
Title: Intercostal Cryoanalgesia for Prevention of Chronic Postoperative Pain Following Video-assisted Thoracoscopic Lung Cancer Resection
Brief Title: Intercostal Cryoanalgesia for Chronic Pain After VATS Lung Resection
Acronym: CRYO-VATS-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-11564
Record Dates: First submitted 2023-05-20; First posted 2023-06-01 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Cryotherapy Effect; Chronic Pain; Lung Cancer; Surgery
MeSH Terms: conditions — Chronic Pain; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Intervention : intercostal cryoanalgesia + single-injection paravertebral block Control group : single-injection paravertebral block
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intercostal cryoanalgesia AND single-injection paravertebral block (Experimental): * Videothoracoscopic-guided single-injection paravertebral block at T5 with 0.4 mL/kg of Bupivacaine 0.5% with adrenalin 5 mcg/mL (maximum 40 mL) at the beginning of surgery
  * Cryoanalgesia 5 cm lateral to the neuraxial, on the inferior costal border, CO2 at (-)50C to (-)70C for 2 minutes, repeated on 7 costal levels (T3-T9), after the lung resection and before chest closure.
  Interventions: Procedure: Cryoanalgesia AND single-injection paravertebral block
- Single-injection paravertebral block (Active Comparator): -Videothoracoscopic-guided single-injection paravertebral block at T5 with 0.4 mL/kg of Bupivacaine 0.5% with adrenalin 5 mcg/mL (maximum 40 mL) at the beginning of surgery
  Interventions: Procedure: Single-injection paravertebral block

INTERVENTIONS:
Procedure: Cryoanalgesia AND single-injection paravertebral block — CO2 Cryoanalgesia AND paravertebral block with Bupivacaine 0.5%
  Arms: Intercostal cryoanalgesia AND single-injection paravertebral block
Procedure: Single-injection paravertebral block — Paravertebral block with Bupivacaine 0.5%
  Arms: Single-injection paravertebral block

SUMMARY:
Intercostal cryoanalgesia is a technique that allows extensive and prolonged analgesia of the hemithorax. The aim of this study is to demonstrate the efficacy of intercostal cryoanalgesia as an adjunct to a single-injection paravertebral block for the prevention of chronic thoracic pain after VATS lung resection surgery.

DETAILED DESCRIPTION:
VATS lung resection is associated with a high incidence of persistent thoracic pain. To our knowledge, there is no study on the effect of cryoanalgesia on the incidence and severity of chronic thoracic pain 3 months after VATS lung resection.

Intercostal cryoanalgesia is a technique that allows extensive and prolonged analgesia of the hemithorax. In a recent study by Ilfeld & al, intercostal cryoanalgesia (combined with a single-injection paravertebral block) was able to drastically lower the incidence of chronic pain after total mastectomy compared to the use of the paravertebral block alone (3% vs 17%).

The aim of this study is to demonstrate the efficacy of intercostal cryoanalgesia for the prevention of chronic thoracic pain after VATS lung resection surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective anatomical pulmonary resection (anatomical segmentectomy, lobectomy or bilobectomy) by VATS for lung cancer
* American Society of Anesthesiologists (ASA) score 1-3

Exclusion Criteria:

* Contraindication to the paravertebral block (coagulopathy, discontinuous paravertebral space, impossible thoracoscopic visualization of the paravertebral space)
* Contraindication to intercostal cryoanalgesia (cold urticaria, cryoglobulinemia)
* Epidural analgesia preferred (high risk of thoracotomy, marginal lung function)
* Surgical criteria (conversion to thoracotomy, non anatomical wedge resection)
* Preoperative thoracic or shoulder pain on the operated side
* Known allergy to acetaminophen, celecoxib, sulfa, or both hydromorphone and morphine
* History of thoracic surgery on the operated site
* Regular use of opioids or medication with effects against neuropathic pain (tricyclics, gabapentinoids, duloxetine, venlafaxine)
* Inability to understand pain scales or to communicate clearly despite adequate teaching
* Contraindication to non-steroidal anti-inflammatory drugs (renal filtration rate < 60 mL/min, active gastric ulcer)
* Pregnancy
* Patient refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
Incidence of persistent thoracic pain | 3 months
  Persistent postoperative thoracic pain (yes or no)

SECONDARY OUTCOMES:
Incidence of persistent thoracic pain | 1 and 6 months
  Persistent postoperative thoracic pain (yes or no)
Severity of persistent thoracic pain | 1,3 and 6 months
  Numerical Rating Scale (NRS) score : scale 0 (no pain) to 10 (worst), at rest and during cough
Incidence of persistent opioid consumption | 1,3 and 6 months
  Persistent postoperative opioid consumption (yes/no)
Incidence of postoperative neuropathic pain | 48 hours, 1 month and 6 months
  DN4 score (10 points) ; positive if 4 points or more
Incidence of new prescription for neuropathic pain medication | 1, 3 and 6 months
  Yes or no
Persistent hypoesthesia over the ipsilateral thorax | 1 and 6 months
  Evaluation of the dermatomal levels of hypoesthesia using a Von Frey monofilament as well as the subjective presence of a sensation of hypoesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Moore, MD, Principal Investigator — Centre Hospitalier de l'Universite de Montreal
Locations (1):
- Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ilfeld BM, Finneran JJ, Swisher MW, Said ET, Gabriel RA, Sztain JF, Khatibi B, Armani A, Trescot A, Donohue MC, Schaar A, Wallace AM. Preoperative Ultrasound-guided Percutaneous Cryoneurolysis for the Treatment of Pain after Mastectomy: A Randomized, Participant- and Observer-masked, Sham-controlled Study. Anesthesiology. 2022 Nov 1;137(5):529-542. doi: 10.1097/ALN.0000000000004334. PMID 35929983